CLINICAL TRIAL: NCT04215510
Title: A Multicenter Randomized Controlled Trial for Comparing Endonasal Surgery and Radiation Therapy (IMRT) for T1-T2 Recurrent Nasopharyngeal Carcinoma
Brief Title: Early Recurrent Nasopharyngeal Cancer: the Effect of Surgery vs IMRT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Principal Investigator, Hongmeng Yu, MD,PhD, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: early-rNPC-RCT-01
Record Dates: First submitted 2019-12-02; First posted 2020-01-02 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
Keywords: endonasal endoscopic surgery; radiation therapy; nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endonasal endoscopic surgery group (Experimental): 143 participants in group 1 will undergo endoscopic surgery
  Interventions: Procedure: endonasal endoscopic surgery
- radiation therapy group (Active Comparator): 143 participants in group 2 will undergo radiation therapy(IMRT)
  Interventions: Radiation: radiation therapy(IMRT)

INTERVENTIONS:
Procedure: endonasal endoscopic surgery — 143 patients will undergo endonasal endoscopic surgery
  Arms: endonasal endoscopic surgery group
Radiation: radiation therapy(IMRT) — 143 patients will undergo radiation therapy.
  Arms: radiation therapy group

SUMMARY:
This study is a multicenter RCT to compare 3-year overall survival(OS) rate, progression free survival(PFS),local progression free survival(LPFS),regional progression free survival(RPFS),distant metastasis free survival(DMFS), and toxicities of endonasal endoscopic surgery versus IMRT.

DETAILED DESCRIPTION:
Local and regional recurrence is a common cause of failure after primary radiotherapy for nasopharyngeal carcinoma. Radiotherapy and surgery are the treatments of choice for recurrent NPC. This study aims to compare 3 year overall survival(OS) rate of surgery versus IMRT.A stratified-block randomized approach will be used to randomly assign patients into two treatment groups after stratification according to N staging (N0 vs non-N0). Patients with rNPC will be recruited and randomized into two groups in 1:1 ratio. The primary outcomes will be 3 year overall survival(OS), the secondary outcome measures will be PFS,LPFS,RPFS,DMFS,and toxicities.Assessment will be performed at baseline and during 3 years post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of recurrent nasopharyngeal carcinoma by pathology or imaging study;
2. Stage T1 or T2 according to AJCC 8th edition ;
3. Aged 18 to 70 years;
4. Without metastasis;
5. previously received 1 course of radiotherapy;
6. Without radiotherapy within 1 year, without local treatment for recurrent disease;
7. Surgical resectable and IMRT suitable;
8. If regional recurrence presented, regional lesion can be treated with local treatments.
9. ECOG score 0 or 1;
10. Sufficient organ function;
11. Acceptable approach of contraception.

Exclusion Criteria:

1. Refuse to sign inform consent;
2. Radiation encephalopathy or leptomeningeal disease (LMD);
3. History of radioactive particle planting;
4. Have uncontrolled intercurrent illnesses which will interfere with the ability to undergo therapy;
5. With prior malignancy (excluding adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer );
6. Any contradiction to surgery;
7. Have any co-existing condition that would preclude full compliance or safety with the study;
8. Presence of a significant neurological or psychiatric disease, including dementia and seizures;
9. Uncontrolled infectious diseases;
10. Female patients who are at pregnancy or lactation.
11. Without personal freedom or independent civil capacity.
12. With serious autoimmune disease.
13. Participants of other interventional clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
3 year Overall Survival (OS) rate | From date of randomization until the date of death from any cause,through study completion,up to 3 years.
  The proportion of patients who survived 3 years

SECONDARY OUTCOMES:
progression free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first，through study completion,up to 3 years.
  the time from randomization to the first recording of disease progression or death from any cause.
Local progression free survival(LPFS) | From randomization to local failure or date of death from any cause,through study completion,up to 3 years.
  the time from randomization to local failure or death
Regional progression free survival(RPFS) | From randomization to regional failure or date of death from any cause, through study completion,up to 3 years.
  From randomization to regional failure or death
Distant metastasis free survival(DMFS) | From randomization to distant metastasis or date of death from any cause, through study completion,up to 3 years.
  From randomization to distant metastasis or death
toxicities | From date of randomization until 3 years after randomization,through study completion,up to 3 years.
  Using CTCAE Version5.0 to evaluate

OTHER OUTCOMES:
quality of life(QoL): EORTC QLQ - H&N35 questionaire | From date of randomization until 3 years after randomization,through study completion,up to 3 years.
  using European Organisation for Research and Treatment of Cancer quality of life questionaire（EORTC QLQ）- H&N35，All of the scales and single-item measures range in score from 0 to 100. For all the scales and single-items a high score represents a high level of symptomatology or problems.
quality of life(QoL): EORTC QLQ - C30 questionaire | From date of randomization until 3 years after randomization,through study completion,up to 3 years.
  using European Organisation for Research and Treatment of Cancer quality of life questionaire（EORTC QLQ) - C30 version3.0. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, MD, Principal Investigator — Eye&ENT Hospital,Fudan University
Locations (3):
- China (3):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Fudan University Shanghai cancer center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No